CLINICAL TRIAL: NCT07272850
Title: Comparison Between Haematological Parameters and Musculoskeletal Ultrasound Findings of Rheumatoid Arthritis Patients Recieving JAK Inhibitors Versus Traditional Treatment
Brief Title: Comparison Between JAK Inhibitors and Traditional Treatment of Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Mohamed Abd Elaal, Lecturer, Assiut University
Other Study IDs: JAK inhibitors in RA
Record Dates: First submitted 2025-10-02; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two groups (1)rheumatoid arthritis receiving JAK inhibitors . (2) rheumatoid arthritis receiving tra
  Interventions: Drug: JAK inhibitors and traditional treatment of rheumatoid arthritis

INTERVENTIONS:
Drug: JAK inhibitors and traditional treatment of rheumatoid arthritis — Type of the study:
  * cross sectional study
  * two groups (1)rheumatoid arthritis receiving JAK inhibitors . (2) rheumatoid arthritis receiving traditional treatement
  2.4. 2- Study Setting: Internal medicine department ,out patient rheumatology clinics of assuit university hospitals 2.4.3- study duration : October 2025 to October 2026
  2.4. 4- Study subjects:
  1. Inclusion criteria:
     * RA patients based on the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classifcation criteria for RA.
     * Age; 18-60
  2. Exclusion criteria:
     * the presence of other autoimmune diseases (e.g., systemic lupus erythematosus or psoriatic arthritis),
     * history of active infections, malignancy, or chronic diseases affecting hematological
     * parameters (e.g., anemia unrelated to RA, chronic kidney disease)
     * RA patients in remission
     * pregnant and lactating female patients
  3. Sample Size Calculation Based on determining the main outcome variable, the estimated

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease that affects about 1% of the world's population [1]. The disease is characterized by synovial membrane inflammation. The impact of RA on quality of life is significant, as it can lead to considerable disability, reduced mobility, and an increased risk of additional health complications [2].

CsDMARDs are the first-line drugs for RA treatment, of which methotrexate (MTX) is the cornerstone drug and monotherapy is recommended as the first choice (3).

However, previous studies had shown that 50% of RA patients had poor treatment effect on methotrexate or inadequate response to re-medication after relapse, resulting in drug resistance (4), resulting in no significant relief of symptoms and still high disease activity. EULAR had indicated that interleukin-6 (IL-6) receptor inhibitors and JAK inhibitors may have advantages over other biological disease-modifying anti-rheumatic drugs (bDMARDs) in patients who were not suitable for csDMARDs (5) Therefore, JAK inhibitors is used as monotherapy or combination therapy, which would provide a new strategy for clinical treatment. A few researches evaluated the relationship between PLT, RBC, Hb, red blood cells-platelet ratio (RPR), and the hemoglobin-platelet ratio (HPR) and RA disease activity. There is growing evidence that metrics like RDW and MPV, as well as the platelet-to-lymphocyte ratio (PLR), neutrophil-to-lymphocyte ratio (NLR), and others have been considered to be accurate, reliable inflammatory biomarkers in autoimmune illnesses[6,7] US has proven itself to be a useful imaging method for assessing articular and periarticular inflammation in small and large joints throughout the last years High resolution musculoskeletal ultrasound (MSUS), incorporating power Doppler ultrasound (PDUS), has demonstrated to be significantly more accurate than clinical evaluation in visualizing the inflammatory process. Furthermore, relatively few studies have examined ankle joint involvement in individuals with RA who lack symptoms [8].

ELIGIBILITY:
Inclusion Criteria:

* • RA patients based on the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classifcation criteria for RA.

  * Age; 18-60

Exclusion Criteria:

* • the presence of other autoimmune diseases (e.g., systemic lupus erythematosus or psoriatic arthritis),

  * history of active infections, malignancy, or chronic diseases affecting hematological
  * parameters (e.g., anemia unrelated to RA, chronic kidney disease)
  * RA patients in remission
  * pregnant and lactating female patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two groups (1)rheumatoid arthritis receiving JAK inhibitors . (2) rheumatoid arthritis receiving traditional treatement
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
changes in hematological parameters as MLR | 1 year
  MLR were determined by dividing the abso- lute neutrophil count by the absolute lymphocyte count, the absolute platelet count by the absolute lymphocyte count, and the absolute monocyte count by the absolute lymphocyte count, respec- tively
improvement in musculoskeletal ultrasound scores. | 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rheumatologyadvisor.com/cch/rheumatoid-arthritis-jak-inhibitors-upadacitinib-tofacitinib-baricitinib/